CLINICAL TRIAL: NCT02961088
Title: Effect of Pasta as Part of Low Glycemic Index Diets on Body Weight and Markers of Adiposity in Humans: A Series of Systematic Reviews and Meta-analyses to Provide Evidence-based Guidance for Nutrition Guidelines Development
Brief Title: Meta-analyses of Pasta as Part of Low Glycemic Index Diets and Adiposity
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: Toronto 3D Knowledge Synthesis and Clinical Trials foundation (Unknown)
Responsible Party: Principal Investigator, John Sievenpiper, Associate Professor, University of Toronto
Other Study IDs: Toronto3D Pasta 2016
Record Dates: First submitted 2016-11-04; First posted 2016-11-10 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes; Prediabetes; Overweight; Obesity; Metabolic Syndrome; Cardiovascular Disease
Keywords: Systematic review and meta-analysis; Evidence-based medicine (EBM); Evidence-based nutrition (EBN); Clinical practice guidelines; Glycemic index; Pasta; Glycemic load; Body weight; Cardiovascular risk factors; Cardiovascular disease
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; Overweight; Obesity; Metabolic Syndrome; Cardiovascular Diseases; Body Weight

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Pasta as part of a low GI/GL diet

SUMMARY:
Pasta is an important example of a food which can lower the glycemic index (GI) of the diet, a property that has been exploited extensively in studies of low GI dietary patterns. Although low-GI dietary patterns have been shown to improve body weight, glycemic control and blood lipids, it is unclear whether pasta as part of low-GI dietary patterns will improve measures of global adiposity including body weight. The lack of high quality knowledge syntheses to support evidence-based dietary guidance of the cardiometabolic benefits of pasta represents an urgent call for stronger evidence. To improve evidence-based guidance for pasta recommendations, the investigators propose to conduct a systematic review and meta-analysis of controlled studies in humans to assess the effect of eating pasta as part of a low GI diet compared to other diets on measures of adiposity (body fatness) in humans. The systematic review process allows the combining of the results from many studies in order to arrive at a pooled estimate, similar to a weighted average, of the true effect. The investigators will be able to explore whether eating pasta as part of a low GI diet has different effects between men and women, in different age groups and in people with high or normal sugar. The findings of this proposed knowledge synthesis will help improve the health of Canadians through informing recommendations for the general public, as well as those at risk of heart disease and diabetes.

DETAILED DESCRIPTION:
Background: Overweight and obesity is a key modifiable risk factor for the prevention and management of type 2 diabetes, dyslipidemia, hypertension, CVD and certain cancers. Low-GI dietary patterns have been shown to improve body weight, among other risk factors including glycemic control and blood lipids, and have been associated with risk reduction of type 2 diabetes and CVD. Current clinical practice guidelines suggest the replacement of high GI foods with low GI foods for improvement of glycemic control and cardiovascular risk factors. Pasta is an important example of a food which can lower the GI of the diet, a property that has been exploited extensively in studies of low GI dietary patterns. However, it is unclear whether pasta as part of low-GI dietary patterns will improve measures of global adiposity, including body weight in addition to other markers of adiposity.

Need for a review: The lack of high quality knowledge syntheses to support evidence-based dietary guidance on pasta represents an urgent call for stronger evidence. A systematic review and meta-analysis of randomized controlled trials remains the "Gold Standard" of evidence to support clinical practice guidelines and public health policy. By pooling the totality of the available evidence, a systematic reviews and meta-analyses of randomized controlled trials would provide the best estimate of the effect of pasta on measures of global adiposity relevant to the prevention and management of overweight and obesity.

Objectives: To provide evidence-based guidance for public health policy, health claims, and nutrition guidelines relating to pasta as part of low GI dietary pattern, the investigators will conduct a systematic review and meta-analysis of randomized controlled trials to assess the effect of past as part of a low GI diet on markers of global adiposity, including body weight in addition to others as well as regional markers of adiposity which have demonstrated clinical relevance.

Design: The planning and conduct of the proposed meta-analyses will follow the Cochrane handbook for systematic reviews of interventions. The reporting will follow the Preferred Reporting Items for Systematic reviews and Meta-Analyses (PRISMA) guidelines.

Data sources: MEDLINE, EMBASE and The Cochrane Central Register of Controlled Trials will be searched using appropriate search terms.

Study selection: Randomized controlled trials that investigate the effect of pasta as part of a low GI dietary pattern on body weight and other markers of adiposity in humans will be included. Trials that are less than 3 weeks diet duration, do not have a control group, include pregnant women, breast feeding women or children, or do not report data on markers of body weight will be excluded.

Data extraction: Two independent investigators will extract information about study design, sample size, subject characteristics, GI/GL diet, follow-up, and the composition of the background diets. Mean ± SEM values will be extracted for all outcomes. Standard computations and imputations will be used to derive missing data. Risk of bias will be assessed using the Cochrane Collaboration risk of bias tool.

Outcome: The primary outcome will be mean differences in body weight as a global marker of adiposity which has demonstrated clinical relevance. Secondary outcomes will be mean differences in other markers of global adiposity with clinical relevance including BMI and percentage body fat, as well as regional markers of adiposity with clinical relevance including waist circumference, waist-to-hip ratio, sagittal abdominal diameter, and visceral adipose tissue [VAT] by imaging modalities.

Data synthesis: Pooled analysis will be conducted using the Generic Inverse Variance method. Separate analyses will be conducted for children and adults. Analyses will be further stratified by metabolic phenotype (normal weight, overweight/obese, metabolic syndrome criteria, diabetes, etc.). Random-effects models will be used even in the absence of statistically significant between-study heterogeneity, as they yield more conservative summary effect estimates in the presence of residual heterogeneity. Fixed-effects models will only be used where there is <5 included studies. Paired analyses will be applied to all crossover trials. Heterogeneity will be tested by the Cochran Q statistic and quantified by the I2 statistic. Sources of heterogeneity will be explored by sensitivity and subgroup analyses. If there are ≥ 10 trial comparisons, then a priori subgroup analyses will also be conducted by dose (<100g/day, ≥100g/day), comparator, follow-up (<6-months, ≥6-months), baseline body weight (BMI ≤25 >25kg/m2), design (parallel, crossover), energy balance (negative, neutral, positive), GI (absolute level [≤55, >55], within-treatment change, between-treatment change), fat intake (absolute level [<30%, ≥30% energy], within-treatment change, between-treatment change), carbohydrate intake (absolute level [<50%, ≥50% energy], within-treatment change, between-treatment change), protein intake (absolute level [<20%, ≥20% energy], within-treatment change, between-treatment change), dietary fibre intake (absolute level [<25g/day, ≥25g/day], within-treatment change, between-treatment change), and risk of bias. Meta-regression will assess the significance of categorical and continuous subgroup analyses. Non-linear relationships will be assessed by spline curve modeling (the MKSPLINE procedure) to assess whether there is a threshold for benefit. If there are ≥10 trial comparisons, then publication bias will be assessed by inspection of funnel plots and the Egger and Begg tests. In the presence of significant publication bias, an adjustment for funnel plot asymmetry will be attempted by using the Duval and Tweedie trim-and-fill method.

Evidence Assessment: The strength of the evidence for each outcome will be assessed using the Grading of Recommendations Assessment, Development and Evaluation (GRADE).

Knowledge translation plan: Results will be disseminated through traditional means such as interactive presentations at local, national, and international scientific meetings and publication in high impact factor journals. Innovative means such as webcasts with e-mail feedback mechanisms will also be used. Knowledge Users will act as knowledge brokers networking among opinion leaders and different adopter groups to increase awareness at each stage. Four Knowledge Users will also participate directly as members of nutrition guidelines committees. Target adopters will include the clinical practice, public health, industry, research communities, and patient groups. Feedback will be incorporated and used to guide analyses and improve key messages at each stage.

Significance: The proposed project will aid in knowledge translation related to the role of pasta as part of a healthy low-GI-dietary pattern on health outcomes strengthening the evidence-base for guidelines and improving health outcomes, by educating healthcare providers and patients, stimulating industry innovation, and guiding future research design.

ELIGIBILITY:
Inclusion Criteria:

* Dietary trials in humans
* Randomized trials
* Trials greater than or equal to 3 weeks duration
* Suitable control group
* Viable outcome data

Exclusion Criteria:

* No assessment of the glycemic index
* Co-intervention present (i.e. the study is designed in such a way that the effect of past as part of a low glycemic index or glycemic load diet can not be isolated)
* Trials looking at the glycemic index of specific foods instead of the diet as a whole
* Trials that did not include pasta as part of the low GI/GL diet
* Trials that included pasta in the control diet
* Trials including pregnant or breast feeding women
* Non-human studies
* Non-randomized trials
* Trials less than 3 weeks duration
* Lack of a suitable control group
* No viable endpoint data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All individuals, with the exception of children and pregnant or breast-feeding women, regardless of health status.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Global measures of adiposity with established clinical relevance - body weight | Up to 20 years
  body weight

SECONDARY OUTCOMES:
Global measures of adiposity with established clinical relevance - BMI | Up to 20 years
  body mass index, BMI
Global measures of adiposity with established clinical relevance - percentage body fat | Up to 20 years
  percentage body fat
Regional measures of adiposity with established clinical relevance - waist circumference | Up to 20 years
  waist circumference
Regional measures of adiposity with established clinical relevance - waist-to-hip ratio | Up to 20 years
  waist-to-hip ratio
Regional measures of adiposity with established clinical relevance - sagittal abdominal diameter | Up to 20 years
  sagittal abdominal diameter
Measures of adiposity by established imaging techniques - visceral adipose tissue [VAT] | Up to 20 years
  visceral adipose tissue [VAT] by imaging modalities

IPD SHARING:
Plan to Share IPD: No
All data will be included in the meta-analyses and available online as supplemental material

REFERENCES:
- [Background] Mirrahimi A, de Souza RJ, Chiavaroli L, Sievenpiper JL, Beyene J, Hanley AJ, Augustin LS, Kendall CW, Jenkins DJ. Associations of glycemic index and load with coronary heart disease events: a systematic review and meta-analysis of prospective cohorts. J Am Heart Assoc. 2012 Oct;1(5):e000752. doi: 10.1161/JAHA.112.000752. Epub 2012 Oct 25. PMID 23316283
- [Background] Turner-McGrievy GM, Jenkins DJ, Barnard ND, Cohen J, Gloede L, Green AA. Decreases in dietary glycemic index are related to weight loss among individuals following therapeutic diets for type 2 diabetes. J Nutr. 2011 Aug;141(8):1469-74. doi: 10.3945/jn.111.140921. Epub 2011 Jun 8. PMID 21653575
- [Background] Larsen TM, Dalskov SM, van Baak M, Jebb SA, Papadaki A, Pfeiffer AF, Martinez JA, Handjieva-Darlenska T, Kunesova M, Pihlsgard M, Stender S, Holst C, Saris WH, Astrup A; Diet, Obesity, and Genes (Diogenes) Project. Diets with high or low protein content and glycemic index for weight-loss maintenance. N Engl J Med. 2010 Nov 25;363(22):2102-13. doi: 10.1056/NEJMoa1007137. PMID 21105792
- [Background] Jenkins DJ, Kendall CW, Augustin LS, Mitchell S, Sahye-Pudaruth S, Blanco Mejia S, Chiavaroli L, Mirrahimi A, Ireland C, Bashyam B, Vidgen E, de Souza RJ, Sievenpiper JL, Coveney J, Leiter LA, Josse RG. Effect of legumes as part of a low glycemic index diet on glycemic control and cardiovascular risk factors in type 2 diabetes mellitus: a randomized controlled trial. Arch Intern Med. 2012 Nov 26;172(21):1653-60. doi: 10.1001/2013.jamainternmed.70. PMID 23089999
- [Derived] Chiavaroli L, Kendall CWC, Braunstein CR, Blanco Mejia S, Leiter LA, Jenkins DJA, Sievenpiper JL. Effect of pasta in the context of low-glycaemic index dietary patterns on body weight and markers of adiposity: a systematic review and meta-analysis of randomised controlled trials in adults. BMJ Open. 2018 Apr 2;8(3):e019438. doi: 10.1136/bmjopen-2017-019438. PMID 29615407